CLINICAL TRIAL: NCT03424499
Title: Randomized Clinical Trial Using Sterile Single-use and Reused Polyvinylchloride Catheter For Intermittent Catheterization With Clean Technique In Neurogenic Bladder Due to Spina Bifida
Brief Title: Sterile Single-use vs Reused Polyvinylchloride Catheter For Intermittent Catheterization In Neurogenic Bladder
Acronym: Catheters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Adrián Gutiérrez González, Dr. med. Adrián Gutiérrez González, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UR16-00005
Record Dates: First submitted 2018-01-23; First posted 2018-02-07 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Neurogenic Bladder Due to Spina Bifida (Disorder)
Keywords: neurogenic bladder; intermittent urethral catheterization; Clean intermittent catheterization
MeSH Terms: conditions — Urinary Bladder, Neurogenic

STUDY DESIGN:
Intervention Model Description: Subjects assigned into 3 parallel groups: Group1 assigned to use a single-use PVC catheter for Intermittent bladder catheterization for neurogenic bladder. Group2 and Group3 will use a reused PVC catheter. Both groups will have a follow-up of 8 weeks. Subjects will be randomized into block sizes of 6 using an electronic list. Both groups will be instructed to use sterile water-soluble lubricant in each catheterization. In the reused catheter group, PVC catheter is washed with water and soap, stored in a container with 0.5% benzalkonium chloride, Group3 catheter washed with water and soap alone. Each catheter is programmed to last a week. Patients/parents are going to be instructed to use clean technique by hand washing with water and soap, and penis/vulva cleansing with antiseptic wipes. Urine cultures will be taken day 0,7,14,28,42 and 56, collecting urine samples from fresh midstream catheter specimen, and evaluation of symptoms related to urinary tract infections.
Who Masked: Outcomes Assessor
Masking Description: Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group A (sterile single-use catheter) Group B (Reused catheter with benzalkonium chloride solution) and Group C (Reused catheter)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single-use catheter (Active Comparator): Participants will use a sterile single-use catheter of polyvinyl chloride (PVC) for intermittent urethral catheterization.
  Intermittent Bladder Catheterization will be done using clean technique, each PVC catheter will be sterile and used only once for each catheterization.
  A Urine culture will be performed at day 0, 7, 14, 28, 49 and 56 (a total of 8 cultures)
  Interventions: Procedure: Single-use catheter; Diagnostic Test: Urine culture
- Reused catheter with 0.5% benzalkonium chloride (Experimental): Participants will use a clean reused catheter of polyvinyl chloride for intermittent urethral catheterization.
  Intermittent Bladder Catheterization will be done using clean technique. The PVC catheter will be used for 1 week, cleaning the catheter with water and soap after each catheterization and stored in a container with 0.5% benzalkonium chloride.
  A Urine culture will be performed at day 0, 7, 14, 28, 49 and 56 (a total of 8 cultures)
  Interventions: Procedure: Reused catheter; Diagnostic Test: Urine culture
- Reused catheter with soap and water (Experimental): Participants will use a clean reused catheter of polyvinyl chloride for intermittent urethral catheterization.
  Intermittent Bladder Catheterization will be done using clean technique. The PVC catheter will be used for 1 week, cleaning the catheter with water and soap after each catheterization.
  A Urine culture will be performed at day 0, 7, 14, 28, 49 and 56 (a total of 8 cultures)
  Interventions: Procedure: Reused catheter; Diagnostic Test: Urine culture

INTERVENTIONS:
Procedure: Single-use catheter — Each urethral catheterization will be done with a new sterile catheter in a period of 8 weeks. Frequency of urethral catheterization will depend of the conditions of each patient (from 3-5 per day). Patients and parents were instructed to use clean technique by hand washing with water and soup, and penis/vulva cleansing with antiseptic wipes. Researchers reinforced the intermittent catheterization technique before the trial.
  Other Names: Single-use catheter intermittent urethral catheterization
  Arms: Single-use catheter
Procedure: Reused catheter — Each catheter is programmed to last 1 week. Evaluation will last a period of 8 weeks. Frequency of urethral catheterization will depend of the conditions of each patient (from 3-5 per day). after catheterization. Each catheter was programmed to last a week. Patients and parents were instructed to use clean technique by hand washing with water and soup, and penis/vulva cleansing with antiseptic wipes. Researchers reinforced the intermittent catheterization technique before the trial.
  Other Names: Reused clean catheter intermittent urethral catheterization
  Arms: Reused catheter with 0.5% benzalkonium chloride; Reused catheter with soap and water
Diagnostic Test: Urine culture — A midstream urine sample will be obtained using sterile catheterization for urine culture performed by health provider. Urine cultures will be done in days 0, 7, 14, 28, 42 and 56.

SUMMARY:
The objective of the study is to determine whether single-use polyvinylchloride (PVC) catheters reduce urinary tract infections (UTI) compared to reused PVC catheters for patients with neurogenic bladder due to spina bifida that require intermittent catheterization for bladder emptying. The investigators conducted a clinical trial with an 8-week follow-up comparing single-use and reused (washed with soap and water, and stored in a container with benzalkonium chloride or washed with soap and water alone) PVC intermittent catheterization. Evaluations were established on days 0, 7, 14, 28, 42, and 56. Participants reported symptoms and urine culture results, collecting urine samples from a fresh midstream catheter specimen using a sterile technique.

DETAILED DESCRIPTION:
The investigators performed a 3-arm clinical trial at the "Dr. José Eleuterio González" University Hospital, a tertiary-care academic hospital in Monterrey, Mexico. The study population were patients from a charity institution for individuals with SB (Asociación de Espina Bífida de Nuevo León A.B.P.) who were treated in our hospital. Patients and parents were offered optional entrance to the study. Inclusion criteria were age ≥ 2 years, diagnosis of SB, self-IC or performed by a trained person, ≥ 3 months using a reused PVC catheter (1 per week) with a clean technique, able to read and understand the informed consent. Exclusion criteria were other causes of NB, symptomatic UTI at the time of initial evaluation (defined as a positive urine culture with pyuria, and odorous urine, flank pain, malaise, or fever), inconsistent IC, an indwelling catheter, allergy to PVC, urethral pathology (eg, stricture, false passage, hypospadias) and rejection to participate in the trial. The use of a prophylactic antibiotic was not an exclusion criterion provided that the participant continued with their usual therapy for the study duration.

The sample size was calculated considering a total of 135 active patients with SB treated in our hospital, using a power of 80%, an expected difference of 50% between arms, and an alpha level set at 0.05. The sample size needed was 75 subjects, using methods for correlated binary data and repeated measures. Subjects were assigned into 3 groups: Group 1 was assigned to use a single-use PVC catheter. Groups 2 and 3 were assigned to use the standard practice modality, a reused PVC catheter. All groups had a follow-up of 8 weeks. Subjects were assigned to block sizes of 6 using a computer-generated list. A blinding process was impossible due to the nature of the intervention.

All groups were instructed to use sterile water-soluble lubricant in each catheterization. In the reused catheter groups, after catheterization, the PVC catheter was washed with water and soap and stored in a container with 0.5% benzalkonium chloride or washed with water and soap alone. Each catheter was programmed to last a week. Patients and parents were instructed to use clean technique by hand washing with water and soap, and penis/vulva cleansing with antiseptic wipes. Researchers reinforced the IC technique before the trial. All participants provided written informed consent.

The primary outcome measure was UTIs. A positive urine culture was defined as the growth of >100,000 CFU. Positive urine cultures were then classified as asymptomatic bacteriuria, defined as a positive urine culture with no symptoms, and UTI, defined as a positive urine culture with cloudy, odorous urine, flank pain, malaise or fever. A total of 6 urine samples were performed per participant, considering baseline the first urine culture, and follow-up the following samples. Participants at baseline were classified as asymptomatic bacteriuria or sterile sample, considering that UTI was an exclusion criterion on baseline sample. Follow-up outcome was classified as sterile (negative urine cultures in all follow-up samples), asymptomatic bacteriuria (at least 1 positive urine culture with no symptoms at any sample), and UTI (at least 1 positive urine culture with symptoms).

The secondary outcomes included person-urine sample UTI, febrile UTI, non-febrile UTI, asymptomatic bacteriuria, and antibiotic use for any reason. Demographics, pharmacologic therapy, urological background, and urodynamic characteristics were evaluated in order to establish an association with the presence of UTI. Urine cultures were programmed at days 0, 7, 14, 28, 42, and 56. Researchers collected all urine samples from a fresh midstream catheter specimen using sterile technique.

An impartial statistician analyzed the data. Categorical variables were expressed in frequencies and percentages. Numerical variables were expressed as means and standard deviation. Clinical and demographic characteristics were analyzed using the χ2 test for categorical variables, and the t-test (or Mann-Whitney test in the absence of normal distribution) for continuous variables. Statistical significance was set at p <0.05. SPSS® software version 20.0 (IBM Corporation, Armonk, NY) was used for all analyses. No funding organization had an influence in the study design, analysis or conclusions.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 2 years,
* diagnosis of spina bifida,
* had self-IC or performed by a trained person ≥ 3 months using reused PVC catheter (1 per week) with clean technique,
* able to read and understand informed consent

Exclusion Criteria:

* other causes of neurogenic bladder,
* symptomatic UTI at the time of initial evaluation,
* inconsistent IC,
* indwelling catheter,
* allergy to PVC,
* urethral pathology (ie stricture, false passage, hypospadias)
* rejection to participate in trial

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
UTIs | Urine cultures were done at day 0, 7, 14, 28, 42, and 56 (8 weeks).
  A positive urine culture is defined as a growth >100,000 CFU of organisms. Positive urine cultures were classified as bacteriuria, defined as a positive urine culture with no symptoms, and UTI, defined as a positive urine culture with cloudy, odorous, flank pain, malaise or fever. A total of 6 urine samples were performed per participant. Outcomes will be measured by Mean and Standard Deviation for UTI, Febrile UTI, Non-febrile UTI and Bacteriuria.

SECONDARY OUTCOMES:
Frequency of bacteriuria and UTI in baseline and follow-up urine cultures. | Urine cultures were done at day 0, 7, 14, 28, 42, and 56 (8 weeks).
  Baseline was considered the first urine culture (day 0), and follow-up the following samples (from day 7 to 56). Participants on baseline were classified as bacteriuria or sterile sample, considering that UTI was an exclusion criterion on baseline sample. Follow-up outcome was classified as sterile (negative urine cultures in all follow-up samples), bacteriuria (at least 1 positive urine culture with no UTI at any sample), and UTI (at least 1 positive urine culture with symptoms).
Comorbidities associated to increased frequency of UTI | Day 0, 7, 14, 28, 42 and 56 (8 weeks).
  Demographic characteristics: gender (frequency and percentage), age in years (mean and standard deviation), and Body Mass Index (weight in kilograms and height in meters will be combined to report BMI in kg/m^2)
  Pharmacologic therapy: The use of antimuscarinic treatment (Frequency and percentage) and antibiotic prophylaxis (Frequency and percentage).
  Urological comorbidities: Bladder diverticula, Vesicoureteral reflux and hydronephrosis (Frequencies and percentages).
  Urodynamic characteristics: hypertonic bladder, overactive detrusor, areflexic bladder, detrusor-sphincter dyssynergy, and filling sensation (Frequencies and percentages).
  This data were evaluated in order to stablish association with the presence of UTI. Clinical and demographic characteristics were analyzed using χ2 test for categorical variables, and T-test (or Mann-Whitney test in the absence of normal distribution) for continuous variables.
Mean person-urine culture UTI, febrile UTI, non-febrile UTI and bacteriuria | Urine cultures were done at day 0, 7, 14, 28, 42, and 56 (8 weeks).
  A positive urine culture is defined as a growth >100,000 CFU of organisms. Positive urine cultures were classified as bacteriuria, defined as a positive urine culture with no symptoms, and UTI, defined as a positive urine culture with cloudy, odorous, flank pain, malaise or fever. A total of 6 urine samples were performed per participant. Outcomes will be measured by Mean and Standard Deviation for UTI, Febrile UTI, Non-febrile UTI and Bacteriuria.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Gutiérrez-González, Principal Investigator — Universidad Autónoma de Nuevo León

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Snow-Lisy DC, Yerkes EB, Cheng EY. Update on Urological Management of Spina Bifida from Prenatal Diagnosis to Adulthood. J Urol. 2015 Aug;194(2):288-96. doi: 10.1016/j.juro.2015.03.107. Epub 2015 Apr 1. PMID 25839383
- [Background] Oakeshott P, Hunt GM, Poulton A, Reid F. Expectation of life and unexpected death in open spina bifida: a 40-year complete, non-selective, longitudinal cohort study. Dev Med Child Neurol. 2010 Aug;52(8):749-53. doi: 10.1111/j.1469-8749.2009.03543.x. Epub 2009 Dec 9. PMID 20015251
- [Background] Lapides J, Diokno AC, Silber SJ, Lowe BS. Clean, intermittent self-catheterization in the treatment of urinary tract disease. J Urol. 1972 Mar;107(3):458-61. doi: 10.1016/s0022-5347(17)61055-3. No abstract available. PMID 5010715
- [Background] Bowman RM, McLone DG, Grant JA, Tomita T, Ito JA. Spina bifida outcome: a 25-year prospective. Pediatr Neurosurg. 2001 Mar;34(3):114-20. doi: 10.1159/000056005. PMID 11359098
- [Background] Guttmann L, Frankel H. The value of intermittent catheterisation in the early management of traumatic paraplegia and tetraplegia. Paraplegia. 1966 Aug;4(2):63-84. doi: 10.1038/sc.1966.7. No abstract available. PMID 5969402
- [Background] Shamout S, Biardeau X, Corcos J, Campeau L. Outcome comparison of different approaches to self-intermittent catheterization in neurogenic patients: a systematic review. Spinal Cord. 2017 Jul;55(7):629-643. doi: 10.1038/sc.2016.192. Epub 2017 Jan 24. PMID 28117329
- [Background] Campbell JB, Moore KN, Voaklander DC, Mix LW. Complications associated with clean intermittent catheterization in children with spina bifida. J Urol. 2004 Jun;171(6 Pt 1):2420-2. doi: 10.1097/01.ju.0000125200.13430.8a. PMID 15126866
- [Background] Schlager TA, Dilks S, Trudell J, Whittam TS, Hendley JO. Bacteriuria in children with neurogenic bladder treated with intermittent catheterization: natural history. J Pediatr. 1995 Mar;126(3):490-6. doi: 10.1016/s0022-3476(95)70477-9. PMID 7869216
- [Background] The prevention and management of urinary tract infections among people with spinal cord injuries. National Institute on Disability and Rehabilitation Research Consensus Statement. January 27-29, 1992. J Am Paraplegia Soc. 1992 Jul;15(3):194-204. doi: 10.1080/01952307.1992.11735873. PMID 1500945
- [Background] Sutherland RS, Kogan BA, Baskin LS, Mevorach RA. Clean intermittent catheterization in boys using the LoFric catheter. J Urol. 1996 Dec;156(6):2041-3. PMID 8911385
- [Background] Moore KN, Burt J, Voaklander DC. Intermittent catheterization in the rehabilitation setting: a comparison of clean and sterile technique. Clin Rehabil. 2006 Jun;20(6):461-8. doi: 10.1191/0269215506cr975oa. PMID 16892928
- [Background] Chaudhry R, Balsara ZR, Madden-Fuentes RJ, Wiener JS, Routh JC, Seed P, Ross SS. Risk Factors Associated With Recurrent Urinary Tract Infection in Neurogenic Bladders Managed by Clean Intermittent Catheterization. Urology. 2017 Apr;102:213-218. doi: 10.1016/j.urology.2016.12.049. Epub 2017 Jan 5. PMID 28065810
- [Background] Mukai S, Shigemura K, Nomi M, Sengoku A, Yamamichi F, Fujisawa M, Arakawa S. Retrospective study for risk factors for febrile UTI in spinal cord injury patients with routine concomitant intermittent catheterization in outpatient settings. Spinal Cord. 2016 Jan;54(1):69-72. doi: 10.1038/sc.2015.170. Epub 2015 Oct 13. PMID 26458969
- [Background] Dean GE. Are Single Use Catheters Worth the Expense? J Urol. 2015 Jul;194(1):12-3. doi: 10.1016/j.juro.2015.04.071. Epub 2015 Apr 16. No abstract available. PMID 25892142
- [Result] Bermingham SL, Hodgkinson S, Wright S, Hayter E, Spinks J, Pellowe C. Intermittent self catheterisation with hydrophilic, gel reservoir, and non-coated catheters: a systematic review and cost effectiveness analysis. BMJ. 2013 Jan 8;346:e8639. doi: 10.1136/bmj.e8639. PMID 23303886
- [Result] Prieto J, Murphy CL, Moore KN, Fader M. Intermittent catheterisation for long-term bladder management. Cochrane Database Syst Rev. 2014 Sep 10;(9):CD006008. doi: 10.1002/14651858.CD006008.pub3. PMID 25208303
- [Result] Pachler J, Frimodt-Moller C. A comparison of prelubricated hydrophilic and non-hydrophilic polyvinyl chloride catheters for urethral catheterization. BJU Int. 1999 May;83(7):767-9. doi: 10.1046/j.1464-410x.1999.00013.x. PMID 10368193
- [Result] Kiddoo D, Sawatzky B, Bascu CD, Dharamsi N, Afshar K, Moore KN. Randomized Crossover Trial of Single Use Hydrophilic Coated vs Multiple Use Polyvinylchloride Catheters for Intermittent Catheterization to Determine Incidence of Urinary Infection. J Urol. 2015 Jul;194(1):174-9. doi: 10.1016/j.juro.2014.12.096. Epub 2015 Jan 10. PMID 25584995
- [Result] Madero-Morales PA, Robles-Torres JI, Vizcarra-Mata G, Guillen-Lozoya AH, Mendoza-Olazaran S, Garza-Gonzalez E, Gutierrez-Gonzalez A. Randomized Clinical Trial Using Sterile Single Use and Reused Polyvinylchloride Catheters for Intermittent Catheterization with a Clean Technique in Spina Bifida Cases: Short-Term Urinary Tract Infection Outcomes. J Urol. 2019 Jul;202(1):153-158. doi: 10.1097/JU.0000000000000244. Epub 2019 Jun 7. PMID 30916625